CLINICAL TRIAL: NCT03970499
Title: Evaluation de l'intérêt de l'élastographie Ultrasonore et du Doppler Ultrasensible peropératoires Dans la Prise en Charge Chirurgicale Des Tumeurs cérébrales
Brief Title: Ultrasound Elastography and Ultrasentive Doppler for Surgery of Brain Tumors
Acronym: ELASTOGLI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PHA017-IZ/ELASTOGLI
Record Dates: First submitted 2019-05-13; First posted 2019-05-31 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Brain Tumor, Primary
Keywords: glioma
MeSH Terms: conditions — Brain Neoplasms; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- glial cerebral tumor (Experimental): patient with an indication of glial cerebral tumor surgery
  Interventions: Procedure: brain tumor resection

INTERVENTIONS:
Procedure: brain tumor resection — Intraoperative brain ultrasound elastography and ultrasensitive doppler during surgery

SUMMARY:
Surgery for brain gliomas is usually guided by different imaging techniques including neuronavigation MRI and intraoperative ultrasound that do not allow visualization of the low-density peri-lesional tumor infiltration present in gliomas and from which the tumor recurs.

Another important aspect in the management of glial tumors is the histological grade. The appearance of new vessels (called neo-angiogenesis) is one of the crucial steps in the life of these tumors, which signifies the transition to anaplasia.

This neoangiogenesis is diagnosed during the anatomopathological analysis of the operative specimen, and may be suspected on preoperative MRI on the so-called infusion sequences.

The objective of this project is to evaluate the potential of two ultrasound modalities - elastography and ultrasensitive Doppler - in helping the surgical management of brain tumors. Ultrasound elastography measures cerebral elasticity and thus indirectly the degree of tumor infiltration; while ultrasensitive Doppler measures intratumoral vascularization, and could therefore help in the diagnosis of tumor anaplasia.

DETAILED DESCRIPTION:
Surgery for brain gliomas is usually guided by different imaging techniques including neuronavigation MRI and intraoperative ultrasound. Unfortunately, MRI and ultrasound do not allow visualization of the low-density peri-lesional tumor infiltration present in gliomas and from which the tumor recurs. Developing tools to identify this "peritumoral" infiltration zone is therefore a major issue in neuro-oncology.

The consistency of brain tumors is a subjective criterion used in cerebral glioma surgery, the tumor area being firmer than the adjacent healthy brain. A pilot study was conducted from December 2012 to March 2014 by the Langevin Institute at La Pitié Salpêtrière. In this study, an intraoperative quantitative measurement of ultrasound elastography was performed on a cohort of patients with brain tumors. A significant difference between elasticity of low grade and high grade gliomas was found. However, in this study, no data on elasticity in a perilational infiltration zone is available.

Another important aspect in the management of glial tumors is the histological grade. The appearance of new vessels (called neo-angiogenesis) is one of the crucial steps in the life of these tumors, which signifies the transition to anaplasia. This neoangiogenesis is diagnosed during the anatomopathological analysis of the operative specimen, and may be suspected on preoperative MRI on the so-called infusion sequences.

The objective of this project is to evaluate the potential of two ultrasound modalities - elastography and ultrasensitive Doppler - in helping the surgical management of brain tumors, through intraoperative ultrasound. Ultrasound elastography measures cerebral elasticity and thus indirectly the degree of tumor infiltration; while ultrasensitive Doppler measures intratumoral vascularization, and can therefore help in the diagnosis of tumor anaplasia.

Ultrasound elastography and ultrasensitive Doppler could enable us to more precisely target the more active tumoral territories (morphological criteria), to better identify the peri-lesional tumor infiltration in order to more precisely guide our resection procedure, and to provide additional information important for pathological analysis.

ELIGIBILITY:
Inclusion Criteria:

* patient with an indication for surgery of a glial cerebral tumor
* informed consent
* age > 18
* social security regime

Exclusion Criteria:

* patient with protection measures as "tutelle or curatelle"
* pregnant woman or woman without contraception measure
* patient under an exclusion period of another research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
ultrasound elastography measurements | 5 minutes, the day of surgery
  Measure of cerebral ultrasound elasticity in three different areas: tumoral, peritumoral, and normal brain (in kPa)
ultrasound ultrasensitive doppler measurements | 5 minutes, the day of surgery
  measurement perfusion by ultrasensitive doppler which consiste to map the power doppler amplitude ( % of vascularization)

SECONDARY OUTCOMES:
Comparaison between ultrasound results and histology | through study completion, an average of 1 year
  histology criteria : type, gradation, neoangiogenesis molecular biology
Correlation between ultrasound results and MRI | through study completion, an average of 1 year
  MRI data : T1, hypersignal FLAIR, regional cerebral blood flow, diffusion
compare elasticity measurements obtained pre-operatively by passive MRI elastography with that obtained intraoperatively by ultrasound elastography. | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ilyess ZEMMOURA, MD PhD, Principal Investigator — CHRU Tours FRANCE
Locations (1):
- Ilyess ZEMMOURA, Tours, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lima GLO, Dezamis E, Corns R, Rigaux-Viode O, Moritz-Gasser S, Roux A, Duffau H, Pallud J. Surgical resection of incidental diffuse gliomas involving eloquent brain areas. Rationale, functional, epileptological and oncological outcomes. Neurochirurgie. 2017 Jun;63(3):250-258. doi: 10.1016/j.neuchi.2016.08.007. Epub 2017 Feb 1. PMID 28161011
- [Result] Mahboob S, McPhillips R, Qiu Z, Jiang Y, Meggs C, Schiavone G, Button T, Desmulliez M, Demore C, Cochran S, Eljamel S. Intraoperative Ultrasound-Guided Resection of Gliomas: A Meta-Analysis and Review of the Literature. World Neurosurg. 2016 Aug;92:255-263. doi: 10.1016/j.wneu.2016.05.007. Epub 2016 May 10. PMID 27178235
- [Result] Ferraro N, Barbarite E, Albert TR, Berchmans E, Shah AH, Bregy A, Ivan ME, Brown T, Komotar RJ. The role of 5-aminolevulinic acid in brain tumor surgery: a systematic review. Neurosurg Rev. 2016 Oct;39(4):545-55. doi: 10.1007/s10143-015-0695-2. Epub 2016 Jan 27. PMID 26815631
- [Result] Coburger J, Merkel A, Scherer M, Schwartz F, Gessler F, Roder C, Pala A, Konig R, Bullinger L, Nagel G, Jungk C, Bisdas S, Nabavi A, Ganslandt O, Seifert V, Tatagiba M, Senft C, Mehdorn M, Unterberg AW, Rossler K, Wirtz CR. Low-grade Glioma Surgery in Intraoperative Magnetic Resonance Imaging: Results of a Multicenter Retrospective Assessment of the German Study Group for Intraoperative Magnetic Resonance Imaging. Neurosurgery. 2016 Jun;78(6):775-86. doi: 10.1227/NEU.0000000000001081. PMID 26516822
- [Result] Gerard IJ, Kersten-Oertel M, Petrecca K, Sirhan D, Hall JA, Collins DL. Brain shift in neuronavigation of brain tumors: A review. Med Image Anal. 2017 Jan;35:403-420. doi: 10.1016/j.media.2016.08.007. Epub 2016 Aug 24. PMID 27585837
- [Result] Chauvet D, Imbault M, Capelle L, Demene C, Mossad M, Karachi C, Boch AL, Gennisson JL, Tanter M. In Vivo Measurement of Brain Tumor Elasticity Using Intraoperative Shear Wave Elastography. Ultraschall Med. 2016 Dec;37(6):584-590. doi: 10.1055/s-0034-1399152. Epub 2015 Apr 15. PMID 25876221